CLINICAL TRIAL: NCT03264846
Title: The Levels of Interleukin-6 and Endocan at Individuals With Polycystic Ovary Syndrome and Periodontal Inflammation
Brief Title: Endocan Levels at Polycystic Ovary Syndrome and Periodontal Inflammation
Status: Completed | Type: Observational
Sponsor: Ebru Saglam (Other)
Collaborators: Ataturk University (Other)
Responsible Party: Sponsor-Investigator, Ebru Saglam, Principal Investigator, Bezmialem Universitesi, Dentistry Faculty, Bezmialem Vakif University
Organization: Bezmialem Vakif University (Other)
Other Study IDs: EbSAGLAM1
Record Dates: First submitted 2017-08-23; First posted 2017-08-29 (Actual); Last update posted 2020-02-10 (Actual); Status verified 2020-02

CONDITIONS: Polycystic Ovary Syndrome; Inflammation Gum; Cytokines
MeSH Terms: conditions — Polycystic Ovary Syndrome; Gingivitis

STUDY DESIGN:
Observational Model: Other | Time Perspective: Cross-Sectional
Patient Registry: Yes
Target Follow-Up Duration: 1 Day
Biospecimen Retention: Samples With DNA — Serum and Saliva
Oversight: Data Monitoring Committee: No | FDA-regulated Drug: No | FDA-regulated Device: No

GROUPS / COHORTS (4):
- Group 1: PCOS participants with periodontitis
  Interventions: Diagnostic Test: Collection of Serum and Saliva Samples
- Group 2: PCOS participants with periodontally healthy
  Interventions: Diagnostic Test: Collection of Serum and Saliva Samples
- Group 3: systemically healthy participants with periodontitis
  Interventions: Diagnostic Test: Collection of Serum and Saliva Samples
- Group 4: systemically and periodontally healthy participants
  Interventions: Diagnostic Test: Collection of Serum and Saliva Samples

INTERVENTIONS:
Diagnostic Test: Collection of Serum and Saliva Samples — Whole saliva samples were obtained via expectorating into polypropylene tubes venous blood were obtained from the antecubital vein via the standard venipuncture method.

SUMMARY:
Periodontal diseases are chronic inflammatory disease occurred by the interaction between pathogenic microorganism and the host defense. Polycystic ovary syndrome (PCOS) is a reproductive and metabolic disease associated with increased risk of cardiovascular events. Endocan is a proteoglycan secreted mainly by endothelial cells under the control of inflammatory cytokines.

Periodontal diseases, including gingivitis, are common chronic infectious diseases caused by predominantly pathogenic microorganisms that colonize the subgingival area and cause local and systemic elevations of proinflammatory cytokines such as Interleukin-6 (IL-6).

Several lines of evidence established the association between periodontal and systemic diseases, including metabolic syndrome, diabetes, and cardiovascular disease.

Because of the fact that both periodontal disease and PCOS are associated with systemic inflammation and insulin resistance, these two disorders may be linked through a common pathophysiologic pathway.

A number of studies have indicated a possible relationship between PCOS and periodontal inflammation. Despite common risk factors, including oxidative stress, the relationship between chronic periodontitis (CP) and PCOS remains unclear.

The aims of the study were to determine serum and saliva Endocan and IL-6 levels and to evaluate the correlation between these two biomarker in women with periodontal disease and PCOS.

ELIGIBILITY:
Inclusion Criteria:

* Newly diagnosed PCOS patients
* Never smokers
* Had no history of systemic disease
* BMI<25 kg/m2
* Participants had ≥20 teeth present.

Exclusion Criteria:

* Pregnancy
* Lactation
* Hemoglobin A1c (HbA1c) ≥ 6.5%
* 2-h oral glucose tolerance test (OGTT-2h) ≥200
* Cushing syndrome, non-classic congenital adrenal hyperplasia, hyperprolactinemia, thyroid dysfunction, and androgen-secreting tumors
* Using antibiotics and antiinflammatory within the past 6 months
* Periodontal treatment within the past 6 months

Ages: 18 Years to 40 Years | Sex: Female | Healthy Volunteers: Yes
Age Groups: Adult
Gender Based: Yes — Only women were included to study.
Study Population: All participants were included among women at the Department of Obstetrics and Gynecology, School of Medicine and Department of Periodontology, Faculty of Dentistry , Ataturk University
Sampling Method: Non-Probability Sample
Enrollment: 87 (Actual)
Dates: Start 2017-04-03 (Actual); Primary Completion 2017-11-29 (Actual); Study Completion 2017-11-29 (Actual)

PRIMARY OUTCOMES:
Serum and salivary Endocan levels | one year
  Enzyme-Linked Immunosorbent Assay (ELISA)
Serum and salivary interleukin-6 levels | one year
  Enzyme-Linked Immunosorbent Assay (ELISA)

SECONDARY OUTCOMES:
Clinical attachment level (CAL) | one year
  Periodontal measurement
Probing pocket depth (PD) | one year
  Periodontal measurement
Gingival Index | One year
  Periodontal measurement

CONTACTS AND LOCATIONS:
Overall Officials: Ebru Sağlam, PhD, Study Director — Bezmialem Vakif University; Ayşe Toraman, Principal Investigator — Ataturk University; Engin Şebin, Principal Investigator — Erzurum Regional Training and Research Hospital; Cenk Fatih Çanakçı, Professor, Study Chair — Ataturk University; Hümeyra Çanakçı, Dr, Principal Investigator — Private Practice; Metin İngeç, Professor, Study Director — Ataturk University
Locations (1):
- Ebru Sağlam, Istanbul, Eyalet/Yerleşke, Turkey (Türkiye)

IPD SHARING:
Plan to Share IPD: Undecided